CLINICAL TRIAL: NCT02192736
Title: Safety and Feasibility Study of Intranasal Mesenchymal Trophic Factor (MTF) for Treatment of Asthma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Translational Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TBS-MTFAS-001
Record Dates: First submitted 2014-07-14; First posted 2014-07-17 (Estimated); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: Asthma
Keywords: asthma; umbilical cord; mesenchymal; stem cells; trophic factors
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Intra-nasal infusion of MTF (Other): Trophic factors from umbilical cord mesenchymal stem cells administered intra-nasally
  Interventions: Biological: Trophic factors from umbilical cord mesenchymal stem cells

INTERVENTIONS:
Biological: Trophic factors from umbilical cord mesenchymal stem cells

SUMMARY:
Allogeneic mesenchymal trophic factors (MTF) from human umbilical cord tissue-derived mesenchymal stem cells (UC-MSC) administered intra-nasally to 20 patients is a safe and useful procedure for inducing improvements in pulmonary function and quality of life in patients with asthma.

DETAILED DESCRIPTION:
The proposed study will assess primary safety and secondary efficacy endpoints of allogeneic UC-MSC-derived MTF administered to patients with asthma. Each patient will receive intra-nasal MTF once per week for a period of 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent form by the subject
* Male or female
* Between 18 and 65 years old and capability to comprehend this trial.
* Asthma diagnosed by a physician at least 1 year prior to study enrollment
* Poorly-controlled asthma at study enrollment. Poorly controlled asthma is defined as: chronic symptoms, episodic exacerbations, persistent and variable airways obstruction despite a continued requirement for short-acting beta 2-agonists despite the use of high doses of inhaled steroids.
* Nonsmokers (stopped smoking at least 1 year ago) and limited life-time history of smoking (less than a 3 pack year history).
* Body mass index 19-40
* On a stable dose of inhaled corticosteroid for at least 4 weeks prior to study entry or had to use a rescue dose during the last 4 weeks.
* FEV1 >50% predicted

Exclusion Criteria:

* Pregnant or lactating women
* Cognitively impaired adults
* Systemic steroids within the 4 weeks prior to enrollment
* Non-steroidal anti-inflammatory drugs (NSAIDs) for arthritis
* Current diagnosis of polyposis or sinusitis.
* Infection treated by antibiotics within the 4 weeks prior to enrollment
* Immunization within the 4 weeks prior to enrollment
* Lung pathology other than asthma
* Other significant non-pulmonary co-morbidities such as: coronary artery disease, peripheral vascular disease, cerebrovascular disease, congestive heart failure with an ejection fraction <50%, liver disease or elevated liver enzymes at baseline, malignancy (excluding non-melanoma skin cancers), AIDS, renal failure with serum creatinine >3.0, or disorders requiring steroid treatment such as vasculitis, lupus, rheumatoid arthritis
* Illicit drug use within the past year
* Current/active upper respiratory infection (URI) (if active URI, wait until asymptomatic for 1 week to enroll)
* Asthma exacerbation within the 4 weeks prior to enrollment (includes ER, urgent care, or hospital visits due to asthma resulting in an increase in asthma-related medications)
* Undergoing evaluation for sleep apnea, or plans to institute treatment for sleep apnea (patients on a stable treatment regimen for sleep apnea for the last 3 months prior to enrollment will be allowed to participate)
* Clinically significant abnormalities present on screening 12-lead electrocardiogram
* Women of childbearing potential using oral contraceptives who are not willing to use a second method of contraception during the study
* Participation in another clinical study within 4 weeks prior to enrollment
* Subject does not sign informed consent

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-07; Primary Completion 2020-04 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Number of patients with adverse events | 1 month
  Evaluated 1 month after the final treatment

SECONDARY OUTCOMES:
Number of patients with a change in pulmonary function from baseline as measured by Forced Expiratory Volume (FEV1) following American Thoracic Society (ATS) guidelines | a) 1 week, 2 weeks, 3 weeks, 4 weeks b) 1 month
  1. After first treatment
  2. After final treatment
Number of patients with a change in pulmonary function from baseline as measured by Forced Vital Capacity (FVC) following American Thoracic Society (ATS) guidelines | a) 1 week, 2 weeks, 3 weeks, 4 weeks b) 1 monrh
  1. After first treatment
  2. After final treatment
Number of patients with a change in quality of life from baseline as measured by the University of Pittsburgh Medical Center (UPMC) Asthma Questionnaire | a) 1 week, 2 weeks, 3 weeks, 4 weeks b) 1 month
  1. After first treatment
  2. After last treatment

CONTACTS AND LOCATIONS:
Overall Officials: Moises Zebede, MD, Principal Investigator — Punta Pacifia Hospital in Panama City, Panama
Locations (1):
- Punta Pacifica Hospital, Panama City, Panama